CLINICAL TRIAL: NCT07386249
Title: Exploration of the Effect of a Wheat Polar Lipid Complex on Vaginal Dryness in Healthy Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seppic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MenoWPLC
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Vaginal Dryness; Menopause Symptoms
Keywords: Menopause; Wheat polar lipids; Vaginal dryness

STUDY DESIGN:
Intervention Model Description: Comparative, randomized, placebo-controlled, double-blind, monocentric interventional study in parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WPLC (Experimental): Dietary supplement - Wheat Polar Lipid Complex
  Interventions: Dietary Supplement: Wheat Polar Lipid Complex
- Placebo (Placebo Comparator): Dietary supplement - Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Wheat Polar Lipid Complex — The study foresees the intake of 1 capsule per day during 12 weeks
  Arms: WPLC
Dietary Supplement: Placebo — The study foresees the intake of 1 capsule per day during 12 weeks
  Arms: Placebo

SUMMARY:
This study aims to explore the positive effect of a dietary supplement composed of wheat polar lipids on vaginal dryness in healthy postmenopausal women

DETAILED DESCRIPTION:
This study is designed as a randomized double-blind placebo-controlled interventional study. One hundred and ten postmenopausal women, aged between 45 and 65 and experiencing vaginal dryness, will be randomly allocated to the control (placebo supplement) or test (active supplement) group. Participants will be supplemented during 12 weeks with those products. Vaginal dryness intensity and menopause symptoms severity will be measured with tests and questionnaires before (baseline), at the middle (6 weeks), and at the end (12 weeks) of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy woman, aged of 45 to 65 years (inclusive)
* In postmenopause, defined according to the STRAW criteria as the absence of menstrual periods for at least 12 consecutive months
* Reporting a vaginal dryness intensity score ≥ 4 on a 0-10 Visual Analogue Scale (VAS), and a score ≥ 16 on the Menopause Rating Scale (MRS)
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Stated willingness to maintain their usual life habits (diet, physical activity, alcohol consumption…)
* Speaking French.

Exclusion Criteria:

* Use of systemic hormonal therapy within the past 3 months
* Use of dietary supplements, herbal products, or over-the-counter remedies intended to alleviate menopausal symptoms within 4 weeks prior to the screening visit (wash-out period ≥ 1 month required)
* Use of vaginal hormonal formulations within 4 weeks prior to screening
* History of hormone-dependent cancers
* History of hysterectomy or bilateral oophorectomy
* Current alcohol dependence or excessive alcohol consumption exceeding an average of 14 standard drinks per week
* Current use of illicit drugs or recent history of drug dependence
* Current or previously diagnosed eating disorders considered likely to impact participant safety or study outcomes
* Presence of severe or uncontrolled chronic medical conditions, or any acute medical condition judged by the investigator to potentially interfere with the MRS assessment or participant safety
* Subject participating in another intervention trial

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological females
Enrollment: 110 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in vaginal dryness intensity | 2, 4, 6, 8, 10 and 12 weeks
  Comparison between groups of the vaginal dryness intensity assessed by a Visual Analogue Scale ranging from 0 ("no dryness at all") to 10 ("extreme vaginal dryness")

SECONDARY OUTCOMES:
Change in vaginal pH level | 6 and 12 weeks
  Comparison between groups of the vaginal pH level assessed using a testing strip
Change in menopausal symptoms severity | 6 and 12 weeks
  Comparison between groups of the menopausal symptoms severity assessed by the Menopause Rating Scale (MRS) questionnaire
Change in menopause-specific quality of life | 6 and 12 weeks
  Comparison between groups of menopause-specific quality of life assessed by the Menopause-Specific Quality of Life (MENQOL) questionnaire
Change in functional and emotional impact of vulvovaginal symptoms | 6 and 12 weeks
  Comparison between groups of functional and emotional impact of vulvovaginal symptoms assessed by the Day-to-day Impact of Vaginal Aging (DIVA) questionnaire
Evolution of self-perceived improvement of vaginal dryness and menopausal symptoms | 6 and 12 weeks
  Comparison between groups of the adjusted for baseline of self-perceived improvement of vaginal dryness and menopausal symptoms assessed by a visual analogue scale, ranging from 0 = not at all to 4 = very much

CONTACTS AND LOCATIONS:
Overall Officials: Louise Deldicque, Pr, Study Director — Université Catholique de Louvain; Sylvie Copine, Dr, Principal Investigator — Université Catholique de Louvain; Laurent Simar, Dr, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Center of Investigation in Clinical Nutrition (CICN), Louvain-la-Neuve, Belgium, Belgium

IPD SHARING:
Plan to Share IPD: No